CLINICAL TRIAL: NCT07059143
Title: A Multicenter Randomized Double-Blind Controlled Trial of Six-Week Transcranial Temporal Interference Stimulation（TIS） Targeting the Right Amygdala for Rapid Alleviation of Depressive Symptoms.
Brief Title: 6 Weeks Right-Amygdala TIS for Depression
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, ZHANG CHENCHEHG, Clinical Neuroscience Center Deputy Director, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025LLSD212-001
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Deep Brain Stimulation; Non-invasive; Amygdala; Temporal Interference; TIS
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amygdala TI (Experimental): 18 sessions will be delivered in 6 weeks: 5 sessions per week for the first two weeks and 2 sessions per week for the following four weeks
  Interventions: Device: Nervio-X
- Controlled TI (Sham Comparator): 18 sessions will be delivered in 6 weeks: 5 sessions per week for the first two weeks and 2 sessions per week for the following four weeks
  Interventions: Device: Nervio-X

INTERVENTIONS:
Device: Nervio-X — An 8-channel TIS device developed by NEURODOME Corporation.

SUMMARY:
The current investigation employs a directed neuromodulation technique, specifically targeting the right amygdala, to ascertain its therapeutic efficacy in managing depressive episodes. The intervention's safety and efficacy will be evaluated using an assessment incorporating depressive symptomatology, cognitive abilities, and daily functions.

ELIGIBILITY:
Inclusion Criteria:

* Age : 18 to 60 years (inclusive), any gender.
* Diagnosis : Major depressive episode diagnosed by study physicians according to the Diagnostic and Statistical Manual of Mental Disorders (5th Edition) (DSM-5), with no restriction on first-onset or recurrent episodes.
* Symptom Severity : 17-item Hamilton Depression Rating Scale (HAMD-17) score ≥ 17 at screening.
* Treatment Stability : Antidepressant regimen must remain unchanged from 30 days prior to signing informed consent through the study duration. Patients using >2 antidepressants or combinations of antidepressant(s) + augmenting agent(s) must be adjusted to ≤2 agents* ≥1 week prior to enrollment.
* Cognitive Capacity : Sufficient literacy and comprehension skills to complete study assessments.
* Compliance : Investigator-confirmed understanding of study objectives/procedures, protocol compliance, and provision of written informed consent.

Exclusion Criteria:

* Comorbidities : Major psychiatric disorders (e.g., schizophrenia, bipolar disorder) Significant neurological conditions (e.g., traumatic brain injury, post-neurosurgical status)
* Medical Devices : Intracranial/cardiac metallic implants or electronic medical devices (e.g., pacemakers, deep brain stimulation systems)
* Recent Interventions : Electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS), or other neuromodulation therapies within 30 days prior to enrollment
* Clinical Instability : Acute suicidality (e.g., active suicidal ideation with intent) Inability to complete study follow-up per investigator judgment
* Concurrent Trials : Participation in other interventional clinical studies during the trial period
* Reproductive Status : Pregnancy, lactation, or plans for conception during the trial
* Suicide Risk : Score ≥3 on Item 3 of the 17-item Hamilton Depression Rating Scale (HAMD-17)
* Any condition deemed to compromise subject safety or study validity per clinical evaluation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology - Self-Report (16-item version) | 6 weeks
  The QIDS-SR16 is a widely used self-report scale for depressive symptoms, containing 16 items that cover all core symptom criteria for DSM-IV major depression. This scale was developed by Rush et al. for rapid assessment of depression symptom severity. Each item has 4 options with a scoring range of 0-3 points, where 0 = no symptoms or mildest symptoms, and 3 = most severe symptoms. The scale demonstrates good internal consistency (Cronbach's α = 0.86) and exhibits high sensitivity for detecting symptom fluctuations.

SECONDARY OUTCOMES:
THINC-it®: An Integrated Tool for Cognitive Dysfunction Screening | Baseline, 2 weeks, 6 weeks, 10 weeks
  THINC-it® is a comprehensive, digitally-based cognitive screening instrument specifically designed to assess cognitive dysfunction in adults with major depressive disorder (MDD). This validated tool comprises five integrated components: four objective cognitive tests (Codebreaker, Trials, Spotter, and SymbolCheck) that evaluate processing speed, executive function, attention, and working memory, plus the PDQ-5-D self-report questionnaire for subjective cognitive assessment. The entire battery requires approximately 10-12 minutes to complete and demonstrates robust psychometric properties with high sensitivity to cognitive changes over time.
Hamilton Depression Rating Scale (17-item version) | Baseline, 1 week, 2 weeks, 6 weeks, 10 weeks
  The Hamilton Depression Rating Scale is a widely utilized clinician-administered instrument for assessing depression severity, consisting of 17 items that evaluate core depressive symptoms. Total scores range from 0-52, with established cutoff points: 0-7 (no depression/remission), 8-13 (mild depression), 14-18 (moderate depression), 19-22 (severe depression), and ≥23 (very severe depression). The HAM-D17 demonstrates good internal consistency reliability with Cronbach's alpha values ranging from 0.747 to 0.829.
Quick Inventory of Depressive Symptomatology - Self-Report (16-item version) | Baseline, 1 week, 2 weeks, 10 weeks
  The QIDS-SR16 is a widely used self-report scale for depressive symptoms, containing 16 items that cover all core symptom criteria for DSM-IV major depression. This scale was developed by Rush et al. for rapid assessment of depression symptom severity. Each item has 4 options with a scoring range of 0-3 points, where 0 = no symptoms or mildest symptoms, and 3 = most severe symptoms. The scale demonstrates good internal consistency (Cronbach's α = 0.86) and exhibits high sensitivity for detecting symptom fluctuations.
Snaith-Hamilton Pleasure Scale (SHAPS) | Baseline, 1 week, 2 weeks, 6 weeks, 10 weeks
  The Snaith-Hamilton Pleasure Scale (SHAPS) is a 14-item self-report instrument designed to assess anhedonia (reduced capacity to experience pleasure) in clinical and research settings. Each item is rated on a 4-point Likert scale (1-4), yielding a total score range of 14-56, where higher scores indicate greater levels of anhedonia. The scale demonstrates excellent internal consistency with Cronbach's alpha values ranging from 0.84 to 0.88 and shows satisfactory test-retest reliability (ICC=0.70).
Hamilton Anxiety Rating Scale (HAMA) | Baseline, 1 week, 2 weeks, 6 weeks, 10 weeks
  The Hamilton Anxiety Rating Scale (HAMA) is a 14-item clinician-administered instrument developed by Hamilton in 1959 to assess anxiety symptom severity in clinical populations. Each item is rated on a 5-point scale (0-4), with total scores ranging from 0-56, where higher scores indicate greater anxiety severity. Score interpretation follows established cutoffs: 0-17 (mild anxiety), 18-24 (mild to moderate anxiety), and 25-30 (moderate to severe anxiety) . The scale demonstrates excellent internal consistency reliability with Cronbach's alpha values consistently ranging from 0.77 to 0.92.
Pittsburgh Sleep Quality Index (PSQI) | Baseline, 2 weeks, 6 weeks, 10 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire designed to assess sleep quality and disturbances over a one-month period. The scale comprises seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each component is scored from 0-3, yielding a global PSQI score ranging from 0-21, where higher scores indicate poorer sleep quality. A global score >5 typically indicates poor sleep quality, while a cutoff of 8 demonstrates optimal sensitivity (0.90) and specificity (0.83) for detecting sleep disturbances. The PSQI demonstrates good psychometric properties with Cronbach's alpha coefficients ranging from 0.64 to 0.89.
36-Item Short Form Health Survey (SF-36) | Baseline and 10 weeks
  The 36-Item Short Form Health Survey (SF-36) is a measure of health-related quality of life consisting of 36 items that assess eight health domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. Items are scored using various response scales (dichotomous, 3-point, 5-point, and 6-point), with domain scores ranging from 0-100, where higher scores indicate better health status. The Cronbach's alpha of the SF-36 ranges from 0.70 to 0.94.
World Health Organization Quality of Life Assessment - Brief Version (WHOQOL-BREF) | Baseline and 10 weeks
  The World Health Organization Quality of Life Assessment - Brief Version (WHOQOL-BREF) is a comprehensive 26-item self-report instrument that evaluates quality of life within the context of an individual's culture, value systems, personal goals, and standards. The scale comprises four domains: Physical Health (7 items), Psychological (6 items), Social Relationships (3 items), and Environment (8 items), plus two additional items assessing overall quality of life and general health. Each item is rated on a 5-point Likert scale, with domain scores transformed to a 0-20 scale or alternatively to a 0-100 scale for standardized comparison. The Cronbach's alpha coefficients of the WHOQOL-BREF ranges from 0.70 to 0.896.

CONTACTS AND LOCATIONS:
Overall Officials: Yiru Fang, MD PhD, Principal Investigator — Ruijin Hospital
Locations (3):
- China (3):
  - The Affiliated Brain Hospital Of Guangzhou Medical University, Guangdong
  - Ruijin Hospital, Shanghai
  - Anding Hospital (Mental Health Center of Tianjin Medical University), Tianjin

IPD SHARING:
Plan to Share IPD: No